CLINICAL TRIAL: NCT03008993
Title: Trial Clinico Controllato e Randomizzato, Con Disegno a Cluster Stepped-wedge, Per Valutare Una Strategia Volta ad Ottimizzare Gli Outcomes Psicosociali in Pazienti Affetti da Cancro
Brief Title: A Stepped Wedge Cluster Randomized Controlled Trial to Assess a Strategy Aiming to Optimize Psychosocial Outcomes in Patients With Cancer
Acronym: HuCare2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Ospitalieri di Cremona (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Parma (Other); Centro di Riferimento Oncologico - Aviano (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other); IRCCS Sacro Cuore Don Calabria di Negrar (Other); Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Principal Investigator, Rodolfo Passalacqua, Head of division, Istituti Ospitalieri di Cremona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HuCare2
Record Dates: First submitted 2016-06-15; First posted 2017-01-04 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Post-Intervention (Experimental): The HQIS comprises three phases: 1) clinician training - to improve communication-relational skills and to instruct on the project; 2) center support - 4 on site visits by experts of the project team, aimed to introduce the project and boost motivation, instruct staff on how to implement recommendations, help with context analysis and identification of solutions; assess actual implementation in the center; 3) implementation of EBM recommendations.
  Interventions: Behavioral: HQIS implementation
- Control (No Intervention)

INTERVENTIONS:
Behavioral: HQIS implementation
  Arms: Post-Intervention

SUMMARY:
INTRODUCTION Our group previously demonstrated the feasibility of the Hucare Quality Improvement Strategy - HQIS, aimed at integrating into practice 6 psychosocial interventions recommended by international guidelines. This randomized trial is designed to assess whether the introduction of the strategy in oncology wards improves patient quality of life.

METHODS AND ANALYSIS This is a multicenter, incomplete stepped-wedge cluster randomized controlled trial, where the intervention strategy is sequentially carried out in three groups of centers (clusters with 5 centers each) and in three equally spaced time periods (epochs) (every 4 months). The study also includes an initial epoch during which none of the centers is exposed to the intervention, and a final epoch when all centers will have implemented the strategy . The intervention is applied at a cluster level (unit of randomization) and assessed at an individual level with cross-sectional model. 720 patients will be included, i.e. 60 patients in each cluster for every detection epoch.

Primary aim is to evaluate the effectiveness of the HQIS vs standard care in terms of improvement of at least one of two domains of HRQoL using the EORTC QLQ-C30 questionnaire, detected at baseline and 3 months after enrolment.

The HQIS comprises three phases: 1) clinician training - to improve communication-relational skills and to instruct on the project; 2) center support - 4 on site visits by experts of the project team, aimed to introduce the project and boost motivation, instruct staff on how to implement recommendations, help with context analysis and identification of solutions; assess actual implementation in the center; 3) implementation of EBM recommendations.

ETHICS AND DISSEMINATION Ethics committee review approval has been obtained from the Ethics Committee of Parma. Results will be disseminated at conferences, in peer-reviewed and professional journals intended for policymakers and managers.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Diagnosis (histological or cytological) of solid tumor communicated to the patient within the previous two months
* About to start a new medical cancer treatment: chemotherapy (IV or oral), molecular target drugs, hormonal therapy, immunotherapy
* Expected survival > 3 months
* Good comprehension of the Italian language
* Who have read, understood, and signed the informed consent.

Exclusion Criteria:

* Previous chemotherapy or other medical cancer treatment
* Recruited in a previous epoch of the study (that is, patients can only participate during one epoch)
* Currently participating in other trials which imply the completion of Patient Reported Outcomes (PROs) in the same period
* Hospitalized
* Currently receiving psychiatric treatment
* Affected by mental or psychiatric disorders, due to cancer or coexisting illness, which interfere with the state of consciousness or impede judgment
* Inability to complete the questionnaire or ensure participation in the three-month follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 762 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) -C30 | baseline - 3rd month
  Quality of life, the primary endpoint of the study, will be assessed with the validated Italian version of the EORTC QLQ-C30 questionnaire, specific for patients with cancer . The tool is self-administered, and comprises 30 questions, 24 of which form nine multi-item scales representing the different aspects, or domains, of QoL: a global health status / QoL scale, five functional scales (physical, role, emotional, cognitive and social), and three symptom scales (fatigue, pain, nausea and vomiting), as well as 6 single items assessing additional symptoms (dyspnoea, loss of appetite, insomnia, constipation, diarrhea) and perceived financial impact of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Passalacqua, Principal Investigator — Istituti Ospitalieri Cremona
Locations (15):
- Italy (15):
  - Azienda USL- Presidio "Di Summa - Perrino", Brindisi
  - Azienda Ospedaliera di Cosenza, Cosenza
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Fano
  - Azienda Ospedaliera Universitaria Policlinico Universitario "G.Martino", Messina
  - IRCCS Istituto Tumori, Milan
  - Azienda Ospedaliera dei Colli, Napoli
  - Azienda Sanitaria Locale, Nuoro
  - Azienda Ospedaliera "P Giaccone", Palermo
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro
  - ASL Ospedale SS Annunziata, Sassari
  - Azienda Ospedaliero Universitaria "San Luigi Gonzaga", Torino
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza, Torino
  - Azienda Ospedaliera Sanitaria Provinciale, Trapani
  - Azienda Ospedaliero-Universitaria di Udine, Udine
  - Ospedale Sacro Cuore "Don Calabria" Presidio ospedaliero accreditato, Verona

REFERENCES:
- [Derived] Caminiti C, Annunziata MA, Verusio C, Pinto C, Airoldi M, Aragona M, Caputo F, Cinieri S, Giordani P, Gori S, Mattioli R, Novello S, Pazzola A, Procopio G, Russo A, Sarobba G, Zerilli F, Diodati F, Iezzi E, Maglietta G, Passalacqua R. Effectiveness of a Psychosocial Care Quality Improvement Strategy to Address Quality of Life in Patients With Cancer: The HuCare2 Stepped-Wedge Cluster Randomized Trial. JAMA Netw Open. 2021 Oct 1;4(10):e2128667. doi: 10.1001/jamanetworkopen.2021.28667. PMID 34648011
- [Derived] Caminiti C, Iezzi E, Passalacqua R. Effectiveness of the HuCare Quality Improvement Strategy on health-related quality of life in patients with cancer: study protocol of a stepped-wedge cluster randomised controlled trial (HuCare2 study). BMJ Open. 2017 Oct 6;7(10):e016347. doi: 10.1136/bmjopen-2017-016347. PMID 28988170